CLINICAL TRIAL: NCT05471999
Title: Small Bowel Perforations: Etiology, Treatment and Outcome
Brief Title: Retrospective Analysis on Small Bowel Perforations
Acronym: SBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 489/2020BO
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-07

CONDITIONS: Small Bowel Perforations
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Retrospective data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with SBP (Other)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — interventional or surgical treatment

SUMMARY:
A retrospective, monocentric, code-related data analysis of patients with small bowel perforations was performed for the period 2010 to 2019.

DETAILED DESCRIPTION:
Analyzed parameters were etiology and timing of perforation, associated morbidity and mortality, type of therapy and its success, and long-term consequences for patients, such as the development of short bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* small bowel perforation in adults

Exclusion Criteria:

* age < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
mortality rate | 30 days
  death by SBP

SECONDARY OUTCOMES:
Small bowel syndrome | 30 days
  malabsorption

CONTACTS AND LOCATIONS:
Overall Officials: S. Bethge, Prof. Dr., Study Chair — Zentrum für klinische Studien der UNiversitätsklinik Tübingen
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Methods would be shared
Supporting Information: Study Protocol
Time Frame: 6 months